CLINICAL TRIAL: NCT00455936
Title: A Randomized Phase III Study of Gefitinib (IRESSATM) Versus Standard Chemotherapy (Gemcitabine Plus Cisplatin) as First-line Treatment for in Never Smokers Advance or Metastatic Adenocarcinoma of Lung
Brief Title: First-line Gefitinib Versus Chemotherapy for Lung Adenocarcinoma in Never Smoker
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Jin Soo Lee, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-126; D7913L00054 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer
Keywords: Adenocarcinoma; NSCLC; gemcitabine; Cisplatin; Gefitinib; Never smoker
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma | interventions — Gefitinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study arm (Experimental): Gefitinib 250mg table/QD, daily every 3 weeks
  Interventions: Drug: Gefitinib
- control arm (Active Comparator): gemcitabine 1250mg/m2 iv on D1 & D8 every 3 weeks Cisplatin 80mg/m2 iv on D1 every 3 weeks
  Interventions: Procedure: chemotherapy

INTERVENTIONS:
Drug: Gefitinib — gefitinib 250mg tablet/ QD daily until Progression
  Other Names: Treamtment Arm
  Arms: study arm
Procedure: chemotherapy — gemcitabine(1250mg/m2 iv on D1 & 8) plus Cisplatin (80mg/m2 iv on D1) every 3 weeks, maximum 9 cycles
  Other Names: standard chemotherapy arm
  Arms: control arm

SUMMARY:
The investigators will conduct the randomized trial to determine the role of Gefitinib monotherapy as first-line setting in adenocarcinoma patients with no history of smoking, as compared with the standard combination chemotherapy.

This is a randomized, open label, parallel group, phase III study in never-smokers with advanced or metastatic adenocarcinoma of lung.

After stratification by gender, performance status, and disease stage, patients will be randomized to one of the two treatment arms to receive either gefitinib or standard chemotherapy until clinical or objective disease progression, unacceptable toxicity or patient's refusal, whichever is sooner. The chemotherapy will be administered for no more than nine cycles.

DETAILED DESCRIPTION:
Gefitinib (Iressa TM) Arm - Gefitinib administration 250mg tablet once daily every 3 weeks

standard chemotherapy arm - gemcitabine (1,250mg/m2 for 30 minutes on day 1 and 8 of a 3 week cycle) plus cisplatin (80mg/m2 on day 1 of a 3 week cycle)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of adenocarcinoma of lung with or without BAC features; however, adenocarcinoma combined with other histology, such as small cell carcinoma or squamous carcinoma, is not allowed.
2. Stage IIIB with malignant pleural effusion/pleural seeding or stage IV patients
3. Age 18-75
4. Never-smoking defined as not more than 100 cigarettes during the lifetime
5. ECOG performance status of 0-2
6. No prior invasive malignancies 5 years prior to study entry except adequately treated cutaneous basal cell carcinoma or uterine cervix in situ cancer
7. Serum creatinine ≤ 1.5 mg/dL, serum bilirubin ≤ 1.2 mg/dL (1 x UNL) and SGOT/SGPT ≤ 100 IU/L (2.5 x UNL)
8. Serum Hgb ≥ 10 gm/dl, platelet count ≥ 100,000/ul, total WBC count >= 4,000/uL, absolute neutrophil count ≥ 1,500/ul
9. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital. The only approved consent form is attached to this protocol
10. The presence of CNS metastases is not considered as an exclusion criterion, provided that there is good control of the symptoms with corticosteroids

Exclusion Criteria:

1. Pregnancy or breast-feeding (women of child-bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy.
2. Major surgery other than biopsy within the past two week.
3. Known severe hypersensitivity to Gefitinib or any of the excipients of this product
4. Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
5. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
6. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
7. Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
8. Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
overall survival | every 12 weeks

SECONDARY OUTCOMES:
To compare Progression-Free survival | every 9 weeks
To compare the quality of life | every 3 weeks
To compare safety profile | every 9 weeks
To collect the tissue samples for the study of predictors of gefitinib (optional) | screening period
To compare the objective response rate (CR+PR) | from the date of randomization to the date of death from any cause the result of each should be recorded separately

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soo Lee, M.D., Study Chair — National Cancer Center, Korea
Locations (3):
- South Korea (3):
  - National Cancer Center, Korea, Goyang-si, Gyenggi-do
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Lee Y, Kim SH, Han JY, Kim HT, Yun T, Lee JS. Early neutrophil-to-lymphocyte ratio reduction as a surrogate marker of prognosis in never smokers with advanced lung adenocarcinoma receiving gefitinib or standard chemotherapy as first-line therapy. J Cancer Res Clin Oncol. 2012 Dec;138(12):2009-16. doi: 10.1007/s00432-012-1281-4. Epub 2012 Jul 7. PMID 22772951